CLINICAL TRIAL: NCT04328181
Title: Comparison of Imaging Quality Between Spectral Photon Counting Computed Tomography (SPCCT) and Dual Energy Computed Tomography (DECT)
Acronym: SPEQUA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL19_0486; ID-RCB (Other: 2019-A02945-52)
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Foot Ulcer; Coronary Artery Disease; Parenchymatous; Pneumonia; Kidney Stone; Inner Ear Disease; Brain Stroke; Joint Diseases; Diabetes; Adrenal Incidentaloma; Hyperaldosteronism; Macroadenoma; Interstitial Lung Disease; Intracranial Arteriovenous Malformations
Keywords: Diagnostic; SPCCT
MeSH Terms: conditions — Diabetic Foot; Coronary Artery Disease; Pneumonia; Kidney Calculi; Labyrinth Diseases; Joint Diseases; Diabetes Mellitus; Adrenal incidentaloma; Hyperaldosteronism; Lung Diseases, Interstitial; Intracranial Arteriovenous Malformations; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPCCT and standard DECT (Experimental): Comparative intra-patients (each patient will have both types of scanner imaging done), clinical superiority study, evaluating the imaging performances (e.g. image quality and radiation dose) of SPCCT and standard DECT for several body regions/anatomical structures.
  Interventions: Device: Spectral Photon Counting Computed Tomography (SPCCT); Device: DECT (Dual Energy CT)

INTERVENTIONS:
Device: Spectral Photon Counting Computed Tomography (SPCCT) — For the dual-layer spectral CT scanner (IQon®, Philips, Amsterdam, The Netherlands), the following parameters will be used for the acquisition:
  * Tube potential 120 kVp;
  * Tube current time product of 150 mAs;
  * Gantry revolution time 0.33 s;
  * Automatic exposure control (angular and longitudinal) combined xyz-axis;
  * Beam collimation geometry 64 x 0.625 mm - scan field-of-view - 22 cm;
Device: DECT (Dual Energy CT) — The SPCCT scanner is a prototype spectral photon-counting computed tomography system derived from a modified clinical CT system with a field-of-view (FOV) of 168 mm in-plane, and a z-coverage of 20 mm. It is equipped with energy-sensitive photon-counting detectors relying on the direct conversion high band gap semiconductor of cadmium zinc telluride (CZT). The electronics comprises 5 rate counters with 5 different configurable energy thresholds. The SPCCT scanner has the following parameters:
  * Base platform : iCT scanner
  * Tube Voltage (kVp) : 120, capability for imaging at 80 and 100 kVp
  * Tube current (mA) : 10 - 300
  * Spatial Resolution : > 30 lp/cm, ≤ 250 µm
  * Z-coverage isocenter (mm) : 20 mm
  * FOV (mm) : 500
  * Minimum rotation time : 0.33 s/rotation
  * Acquisition modes : Axial, Helical, Step & Shoot

SUMMARY:
This pilot study wants to determine to which extent SPCCT allows obtaining images with improved quality and diagnostic confidence when compared to standard Dual Energy CT (DECT), both with and without contrast agent injection.

Depending on the anatomical structures/organs to be visualized during CT examinations, different scanning protocols are performed with quite variable ionizing radiation doses. Therefore, in order to obtain the most extensive and representative results of the improvement in image quality between SPCCT and DECT that will be performed CT imaging on several body regions and structures, including diabetic foot, diabetic calcium coronary scoring, adrenal glands, coronary arteries, lung parenchyma, kidney stones, inner ear, brain and joints, earl/temporal bone, colorectal carcinosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting following one of following medical conditions:

  1. Asymptomatic type 1 or 2 diabetes as regard to cardiovascular risks
  2. Diabetic foot ulcer
  3. Adrenal glands lesions: Adrenal incidentaloma or hyperaldosteronism or macroadenoma
  4. Urinary stone(s)
  5. Known Coronary artery disease: Stent imaging or control of calcified plaques
  6. Diffuse Interstitial Lung Diseases: Idiopathic Pulmonary Fibrosis, Hypersensitivity Pneumonitis, Ground Glass Opacification, Chronic Thromboembolic Pulmonary Hypertension
  7. Conductive hearing loss
  8. Brain stroke (late or post thrombectomy)
  9. Intracranial arteriovenous malformation treated with coils or Onyx
  10. Joints diseases in haemophilia
  11. Ear/temporal bone
  12. Colorectal carcinosis
  13. Dissection aortique de type A opérée ou de type B non opérée, hématome intramural
* Patient has accepted to participate to the study and has signed the written consent;
* Pre-menopausal women only: Negative urinary pregnancy test on the day of imaging before the administration of study drug;
* Patient is affiliated to the French social security

Exclusion Criteria:

* Contraindication to the use of iodine containing contrast media (including subjects with suspicion for/or known to have NSF) (if injection);
* History of severe allergic or anaphylactic reaction to any allergen including drugs and contrast agents (as judged by the investigator, taking into account the intensity of the event);
* History of delayed major or delayed cutaneous reaction to Iomeron injection
* Estimated Glomerular Filtration Rate (eGFR) value < 30 mL/min/1.73 m2 derived from a serum creatinine result within 1 month before the imaging for examinations with contrast agent.
* Any subject on hemodialysis or peritoneal dialysis;
* Suspected clinical instability or unpredictability of the clinical course during the study period (e.g. due to previous surgery);
* Pregnant or nursing (including pumping for storage and feeding);
* Patient under guardianship, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
quality of the images | Day 8
  A single four-point scale will be used (1: unacceptable, 2: usable under limited conditions, 3: probably acceptable, 4: fully acceptable) based on the European guidelines on quality criteria for computed tomography

SECONDARY OUTCOMES:
Diagnostic confidence graded | Day 8
  The diagnostic confidence grade will be calculated on a four-point scale (1: insufficient, 2: poor, 3: average, 4: good).
Subjective image quality graded | Day 8
  It will be calculated on a five-point scale (1: poor, 2: fair, 3: average, 4: good, 5: excellent) for each following criterion: noise, artifacts and sharpness.
CT Dose Index volumic (CTDIvol) | Day 8
  To determine the radiation dose delivered to the patients during the DECT and SPCCT imaging procedures.
  The CTDI is an estimation of the dose delivered to the organs for each acquired section that is based on acquisition parameters of a water phantom with a 32 cm diameter. The value is expressed in milligray (mGy).
Dose Length Product (DLP) | Day 8
  To determine the radiation dose delivered to the patients during the DECT and SPCCT imaging procedures.
  The DLP is obtained as follows: CTDI * length of body explored = value in mGy.cm.
Equivalent dose (mSv) | Day 8
  To determine the radiation dose delivered to the patients during the DECT and SPCCT imaging procedures.
  The equivalent dose is obtained by multiplying the DLP to the specific organ conversion factor.
Quantitatively image quality : Noise | Day 8
  The noise by selecting regions of interest (ROI) will calculated.
Quantitatively image quality : Density | Day 8
  The density (HU) by selecting regions of interest (ROI) will calculated.
Quantitatively image quality : contrast-to-noise ratio | Day 8
  The contrast-to-noise ratio (CNR) by selecting regions of interest (ROI) will calculated.
Depiction of anatomical structures of interest | Day 8
  Depiction of anatomical structures of interest will be graded on a four-point scale (1: visualization just possible, 2: unclear borders but different structures already visible, 3: very good visualization, well-defined anatomy, 4: perfect delineation of anatomy).
Radiation dose | Day 8
  An average radiation dose delivered to the patients for each clinical application will be calculated.
Statistical comparison between SPCCT and DECT | Day 8
  Statistical comparison between SPCCT and DECT will be performed over all images and anatomical structures globally and also for each clinical application of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DOUEK, Pr, Principal Investigator — Service de Radiologie, l'Hôpital Louis Pradel - Hospices Civils de Lyon
Locations (1):
- Hôpital Cardiologique Louis Pradel - Hospices Civils de Lyon, Bron, Avenue Doyen Lépine, France